CLINICAL TRIAL: NCT06107049
Title: Probiotics Improve Sleep Quality: a Randomized Placebo-controlled Trial
Brief Title: the Effect of Probiotic on Sleep Quality Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2023006
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Poor Quality Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Participants in the probiotic group received 3g of BLa80 product per day.
  Interventions: Dietary Supplement: BLa80
- Placebo group (Placebo Comparator): Participants in the placebo group received 3g of maltodextrin per day.
  Interventions: Dietary Supplement: BLa80

INTERVENTIONS:
Dietary Supplement: BLa80 — During the experiment, the subjects took a packet of probiotics every day, and the sleep condition, anxiety level and memory level of the subjects were evaluated by questionnaires and ability tests. The questionnaire included PSQI Pittsburgh Sleep Quality Index scale, ISI Insomnia Severity Index Scale and GSRS gastrointestinal symptom Score scale.

SUMMARY:
The goal of this clinical trial is to learn about the improvement of sleep quality of probiotic BLa 80 in 110 healthy college students. The main question it aims to answer is whether probiotic BLa80 can effectively improve the sleep quality of college students. The experiment commenced with participants continuously consuming the recommended amount of the probiotic powder for approximately 8 weeks. Simultaneously, they were required to fill out an "Effect Evaluation Form" every week and submit it to relevant department. At the end of the first and eighth weeks, participants underwent tests for five liver functions, four lipid profiles, blood sugar, and uric acid levels, as well as stool sample collection. They then completed the "Mid-Term Effect Evaluation Form".

DETAILED DESCRIPTION:
Over the past few decades, the health benefits of probiotics have garnered extensive scientific attention. Particularly in the treatment of gastrointestinal and metabolic disorders, probiotics have shown potential therapeutic effects. The benefits of probiotics to the intestinal environment include improving intestinal barrier function, producing antimicrobial substances, competing with pathogenic bacteria, and regulating cavity acidity. However, research results on the benefits of probiotics for healthy adults are inconsistent. This may be due to variations in consumer sensitivity to the effects of probiotics and differences between probiotic products. The relationship between gut microbiota and human health has been widely recognized, especially in relation to diseases like obesity and diabetes. To verify the effects of the Bifidobacterium BLa80 product, a consumer test experiment was conducted, aiming to test and collect data on the changes in the gut microbiota of participants before and after using the product. The test plan lasted for 10 weeks, including a washout period at the beginning and end. During the experiment, participants consumed Bifidobacterium BLa80 and underwent multiple health checks and evaluations.

ELIGIBILITY:
Inclusion Criteria:

* PSQI Pittsburgh Sleep Quality Index score > 6 and < 18;
* ISI insomnia Severity Index score > 8 and < 23.

Exclusion Criteria:

* Those who have been diagnosed with diabetes or have high blood sugar are not recommended to participate in the test;
* Mental or nervous system diseases, celiac disease, lactose intolerance, allergy;
* Have the following diseases: irritable bowel syndrome, diabetes, ulcerative colitis, etc.;
* Recent antibiotic treatment (i.e. < 3 months before study start);
* Participants who smoked more than 10 cigarettes per day were excluded;
* Other people with special circumstances are not recommended to participate, such as those who are allergic to probiotic products;
* Pregnant women, breastfeeding women and people under 19 years old and over 45 years old should not be tested.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in sleep quality | 8 weeks
  ISI insomnia Severity Index Scale questionnaire（It is divided into 7 items, with a total score of 28 points. 0 to 7 is divided into clinically insignificant insomnia, 8 to 14 is divided into mild insomnia, 15 to 21 is divided into moderate insomnia, and 22 to 28 is divided into severe insomnia.）

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Technology, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No